CLINICAL TRIAL: NCT06802419
Title: A Comparative Study Between the Effect of Continuous Adductor Canal Block Versus Continuous Adductor Canal Block With Additional Infiltration Between The Popliteal Artery and Capsule of The Knee (IPACK) After Arthroscopic Knee Surgeries
Brief Title: Effect of Continuous Adductor Canal Block Versus Continuous Adductor Canal Block With Additional Infiltration Between The Popliteal Artery and Capsule of The Knee (IPACK) After Arthroscopic Knee Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nada Ezzat, Assistant Lecturer of Anesthesiology, Intensive Care and Pain Medicine, Faculty of Medicine, Ain shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD134/2024
Record Dates: First submitted 2025-01-21; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Continuous Adductor Canal Block; Infiltration Between The Popliteal Artery and Capsule of The Knee; Arthroscopic Knee Surgeries
MeSH Terms: interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Patients will receive continuous adductor canal block.
  Interventions: Other: Continuous adductor canal block
- Group 2 (Experimental): Patients will receive Continuous Adductor Canal Block with additional Infiltration between The Popliteal Artery and Capsule of The Knee
  Interventions: Other: Continuous Adductor Canal Block with additional Infiltration between The Popliteal Artery and Capsule

INTERVENTIONS:
Other: Continuous adductor canal block — Patients will receive continuous adductor canal block.
  Arms: Group 1
Other: Continuous Adductor Canal Block with additional Infiltration between The Popliteal Artery and Capsule — Patients will receive Continuous Adductor Canal Block with additional Infiltration between The Popliteal Artery and Capsule of The Knee
  Arms: Group 2

SUMMARY:
This study aims to evaluate the effect of Continuous Adductor Canal Block only versus adding posterior knee block, known as the Infiltration between the Popliteal Artery and Capsule of the Knee (IPACK) block with Continuous Adductor Canal Block (CACB) after arthroscopic knee surgeries.

DETAILED DESCRIPTION:
Enhanced recovery after arthroscopic knee surgery is gaining popularity in orthopedic surgeries. Motor preservation with adequate analgesia has become the optimal postoperative goal, enabling earlier physical therapy, faster recovery, and early hospital discharge. Spinal anesthesia for knee arthroscopy has favorable outcome effects compared with general anesthesia. The positive physiological effects of the provided sympathetic blockade with less blood loss, increased leg blood flow, and better initial pain relief explain this.

An ideal nerve block that targets the sensory nerves and spares the motor function can facilitate early ambulation and rehabilitation, a major goal for patients undergoing arthroscopic knee surgery.

A novel technique for posterior knee block, known as the infiltration between the popliteal artery and capsule of the knee (IPACK) block combined with continuous adductor canal block (CACB) would reduce opioid requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 65 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) Physical Status Class I to II.
* Patients with successful spinal anesthesia.
* Patients scheduled for elective arthroscopic knee surgery for anterior cruciate ligament (ACL) and posterior cruciate ligament (PCL) repair.

Exclusion Criteria:

* Declining to give written informed consent.
* History of allergy to the medications used in the study.
* Contraindications to regional anesthesia (including coagulopathy and local infection).
* Polytrauma patients having lower limb fractures.
* Patients with pre-existing myopathy or neuropathy on the operating limb.
* Patients with diabetes mellitus.
* Psychiatric disorder.
* Morbid obesity [body mass index (BMI) > 45kg/m2].
* Complicated Surgery.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  The degree of pain will be assessed using the Visual Analogue Scale (VAS). VAS score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. No pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).

SECONDARY OUTCOMES:
Total Nalbuphine consumption | 24 hours postoperatively
  Rescue analgesia will be given when VAS score ≥ 30 mm, in the form of IV injection of 10 mg Nalbuphine. Followed by reassessment of pain after 10 minutes, a second dose of Nalbuphine will be given if still VAS score ≥ 30 mm.
Straight leg rise | 24 hours postoperatively
  Straight leg rise (SLR) will be recorded.
Range of motion | 24 hours postoperatively
  Range of motion (ROM) will be recorded
Rate of complications | 24 hours postoperatively
  Rate of complications like falling will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.